CLINICAL TRIAL: NCT00627419
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study Evaluating the Safety and Antitumor Activity of IPI-504, A Novel Small Molecule Inhibitor of Heat Shock Protein 90 (HSP90), in Patients With Metastatic Melanoma
Brief Title: A Study Evaluating the Safety and Antitumor Activity of IPI-504, in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed & recruitment will not recommence
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP159
Record Dates: First submitted 2008-02-21; First posted 2008-03-03 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): IPI-504
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — Dose as a 30 to 60 minute IV infusion as part of a 21-day treatment cycle until unacceptable toxicity, disease progression, initiation of alternative anticancer therapy, or other reasons for patient withdrawal. IPI-504 will be administered twice weekly on Study Days 1, 4, 8, and 11 of each 21-day cycle.

SUMMARY:
To evaluate the antitumor activity of IPI-504 in patients with metastatic melanoma.

DETAILED DESCRIPTION:
To evaluate the antitumor activity of IPI-504 in patients with metastatic melanoma and to assessment of antitumor activity is the 6-month progression-free rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable, Stage IV or recurrent melanoma, including mucosal melanoma (based on American Joint Committee on Cancer [AJCC] staging [Balch, 2001], see Appendix A).
* Prior therapy with chemotherapy and/or immunotherapy for melanoma is allowed provided that therapy ended prior to study entry and all treatment-related toxicities have resolved to NCI CTCAE Grade ≤ 1 or patient's baseline;
* Measurable disease (based on RECIST [Therasse, 2000]) defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan;
* Have melanoma that can be biopsied once prior to treatment (all patients), and a second time during treatment with IPI504 (stage 2 patients);
* Willingness for tumor biopsy at screening (all patients) and once during treatment (stage 2 patients only);
* Males and females of at least 18 years of age at the time of study entry;
* Female patients must be of non child-bearing potential (defined as being >1 year post-menopausal) or using effective contraception, eg, use of oral contraceptives with an additional barrier method (since the study drug may impair the effectiveness of oral contraceptives), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, or total abstinence, from the time the informed consent is signed through 30 days after the last dose of IPI-504. Male patients must be surgically sterile or use a double-barrier method of contraception (condom with spermicide) from the time of the initiation of IPI-504 through 30 days after the last dose of IPI-504;
* Eastern Cooperative Oncology Group performance status of 0 to 2;
* Life expectancy of at least 16 weeks;
* White blood cell (WBC) count ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥ 100,000/mm3; Prothrombin time or international normalized ratio within normal range (unless a patient is receiving anticoagulation therapy), or PTT within normal range;
* Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (by Cockroft-Gault method);
* Total bilirubin ≤ 1.5 × ULN [unless due to Gilbert's syndrome (unconjugated hyperbilirubinemia) in which case the total bilirubin should be ≤ 3.5 mg/dL], AST and ALT ≤ 2.5 × ULN, hepatic alkaline phosphatase ≤ 2.5× ULN;
* LDH ≤ 1.5 × ULN;
* Patients who have had prior radiation therapy are eligible provided that therapy was palliative in nature, not in the area where the tumor will be biopsied, at least one measurable lesion outside the radiation field, and all radiation-related toxicities have resolved to NCI CTCAE Grade ≤ 1 or patient's baseline;
* Patients who had recovered from prior major surgery are eligible if all surgical wounds have healed;
* Written informed consent and HIPAA authorization obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Received an investigational agent or therapy with any other kinase inhibitor within 2 weeks prior to study entry or any other antitumor therapy, such as cytostatic and/or cytotoxic drugs, hormonal therapy, radiation therapy, immunotherapy, or any biological response modifiers within 4 weeks prior to study entry;
* Previous treatment with 17-AAG, 17-dimethylaminoethylamino-17-demethoxygel-danamycin (17-DMAG), or other known Hsp90 inhibitor;
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer;
* Current or planned participation (from the day of study entry through 30 days after the last dose of IPI-504) in a research protocol in which an investigational agent or therapy may be administered;
* Initiation or discontinuation of concurrent medication that alters CYP3A activity (see Appendix C) within 2 weeks prior to treatment with IPI-504. Patients who are on a stable dose of drugs known to alter CYP3A activity for > 2 weeks are eligible to enroll;
* Presence of active infection or systemic use of antimicrobials within 72 hours prior to treatment with IPI-504;
* Known brain metastases or primary brain tumors. Patients with ≤ 2 lesions are eligible provided:

  * Treated with surgery or stereotactic radiosurgery
  * The lesions are < 3 cm in size and have been stable for 2 months (by CT/MRI)
  * The patient has been off steroids for at least 1 week prior to dosing and:
  * The patient is allowed to have had whole brain radiation if performed in conjunction with surgery/stereotactic radiotherapy and the last dose of radiation occurred at least 2 months prior to dosing with IPI504.
* Significant comorbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study (eg, cardiac disease such as acute coronary syndrome or unstable angina within 6 months, uncontrolled hypertension, cirrhotic liver disease, cerebrovascular accident, or other conditions);
* History of prior malignancies within the past 5 years other than non-melanomatous skin cancers that have been controlled, carcinoma in situ of the cervix, T1a or b prostate cancer noted incidentally during a transurethral resection of prostate (TURP) with prostate-specific antigen values within normal limits since TURP, or superficial bladder cancer;
* Women who are pregnant or lactating;
* Sinus bradycardia (resting heart rate < 50 beats/min) secondary to intrinsic conduction system disease; Patients with sinus bradycardia secondary to pharmacologic treatment may enroll if withdrawal of the treatment results in normalization of the resting heart rate to within normal limits;
* Screening QTc > 450 msec in males; QTc > 470 msec in females, or previous history of QTc prolongation while taking other medications; or
* Active or recent history (within 3 months) of keratitis or keratoconjunctivitis, confirmed by ophthalmology or optometry exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluating the antitumor activity of IPI-504 in patients with metastatic melanoma. The primary assessment of antitumor activity is the 6-month progression-free rate. | from the first administration of IPI-504 through 30 days after the last dose of IPI-504

SECONDARY OUTCOMES:
Evaluating other antitumor activities, safety, and PK parameters of IPI-504 in this patient population. | from the first administration of IPI-504 through 30 days after the last dose of IPI-504 (confirm)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Santabarbara, M.D., Study Director — Infinity Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Arizona Cancer Center, Tuscon, Arizona
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana Univ. Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Comprehensive Cancer Center, Rochester, Minnesota
  - Washington School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Univ. of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Univ. of TX, MD Anderson Cancer Center, Houston, Texas